CLINICAL TRIAL: NCT03847805
Title: Effectiveness of a Program of Scapulothoracic and Glenohumeral Stabilization Exercises in Boulderers. A Randomized Pilot Study.
Brief Title: Scapulothoracic and Glenohumeral Stabilization Exercises in Boulderers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Real Fundación Victoria Eugenia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EJERESC
Record Dates: First submitted 2019-02-19; First posted 2019-02-20 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Sports Physical Therapy
Keywords: Bouldering; Exercise; Shoulder; Stability; Performance
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The experimental group followed a program that included three scapulothoracic stabilization exercises and three for glenohumeral stability, while subjects in the control group only performed the glenohumeral stabilization exercises. Two weekly sessions were carried out over a period of 6 weeks, and each session lasted 30 minutes. The intervention was conducted before starting the training session, to avoid muscle fatigue.
  Interventions: Other: Scapulothoracic and glenohumeral stabilization exercises
- Control (Active Comparator): The control group followed a program of glenohumeral stabilization exercises,
  Interventions: Other: Glenohumeral stability exercises

INTERVENTIONS:
Other: Scapulothoracic and glenohumeral stabilization exercises — The experimental group followed a program that included three scapulothoracic stabilization exercises and three for glenohumeral stability, while subjects in the control group only performed the glenohumeral stabilization exercises. Two weekly sessions were carried out over a period of 6 weeks, and each session lasted 30 minutes. The intervention was conducted before starting the training session, to avoid muscle fatigue. Three series, with 10 repetitions of each exercise, with one minute rest between series.
  Other Names: Scapulothoracic stabilization
  Arms: Experimental
Other: Glenohumeral stability exercises — the control group only performed the glenohumeral stabilization exercises. Two weekly sessions were carried out over a period of 6 weeks, and each session lasted 30 minutes. The intervention was conducted before starting the training session, to avoid muscle fatigue.
  Other Names: Glenohumeral stabilization
  Arms: Control

SUMMARY:
Introduction. In the block climbing, the fluidity with which the athlete climbs a certain route is fundamental. The speed with which the movements are executed and the number of grippers of upper limbs is related to sports performance. Shoulder injuries are very prevalent in this sport. The inhibition of the stabilizing musculature can alter joint positioning and its normal biomechanics.

Objective. To evaluate the efficacy of a program of stability exercises, scapulothoracic and glenohumeral, in the improvement of shoulder stability and sports performance, in boulder climbers.

Material and method. Forty randomized subjects will be recruit into two groups: experimental (scapulothoracic and glenohumeral stability exercises) and control (glenohumeral stabilization). The stability of the shoulder (Closed Kinetic Chain Upper Extremity Stability Test) and the sports performance (Climbing Test) will be evaluated. The intervention last 6 weeks, with two weekly sessions of 30 minutes each. Differences between evaluations will be analyzed with the t-sudent for related samples and the intra- and intersubject effect with the repeated measures ANOVA test.

ELIGIBILITY:
Inclusion Criteria:

* Being climbers
* Between the ages of 18 and 40 years
* Belonging to the Boulder Madrid Climbing Gym
* Who climbed at least twice a week
* Having at least 6 months of experience

Exclusion Criteria:

* Were participating in competitions at the time
* Presented pathologies of the upper limb
* Used any type of ergogenic aid
* Had not signed the informed consent document.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-03-20 (Estimated); Study Completion 2019-04-20 (Estimated)

PRIMARY OUTCOMES:
Change from baseline stability of the shoulder after treatment and at 6 weeks | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The investigators used the Closed Kinetic Chain Upper Extremity Stability Test (CKCUEST). This scale evaluates the number of upper limb movements the subject is able to make during 15 seconds. A higher score represents better shoulder stability.

SECONDARY OUTCOMES:
Change from baseline time need to complete a given climbing route and number of grips during climbing after treatment and at 6 weeks | Screening visit, within the first seven days after treatment and after one month follow-up visit
  Bouldering test, replicating the demands of a competition. The test was carried out on a 4-meter-high wall and with a 20 degree inclination, having a route with 15 climbing holds: 3 small, 7 medium and 5 large. A start hold and an end hold were clearly identified. The climber had 5 minutes to visualize the route, in a familiarization process often used in competitions. Before the test participants was told that they should be as efficient as possible in their movements. The time taken by the climber to complete the route was recorded, and the number of grips for the route.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Study Director — Universidad Europea de Madrid
Locations (1):
- Real Fundación Victoria Eugenia, Madrid, Spain